CLINICAL TRIAL: NCT00601107
Title: A Multicenter, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Assess the Efficacy and Safety of Doxercalciferol Capsules in the Treatment of Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Safety and Effectiveness of Doxercalciferol Capsules in Participants With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HECTPS02507
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
Keywords: psoriasis; psoriasis vulgaris; plaque psoriasis; chronic plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — 1 alpha-hydroxyergocalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Doxercalciferol 2.5 mcg/day (Experimental): Doxercalciferol 2.5 microgram (mcg) capsule orally once daily up to Week 24.
  Interventions: Drug: Doxercalciferol
- Doxercalciferol 5 mcg/day (Experimental): Doxercalciferol 5 mcg capsules orally once daily up to Week 24.
  Interventions: Drug: Doxercalciferol
- Doxercalciferol 7.5 mcg/day (Experimental): Doxercalciferol 7.5 mcg capsules orally once daily up to Week 24.
  Interventions: Drug: Doxercalciferol
- Placebo (Placebo Comparator): Placebo matching to doxercalciferol capsules orally once daily up to Week 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxercalciferol
  Other Names: Hectorol®
  Arms: Doxercalciferol 2.5 mcg/day; Doxercalciferol 5 mcg/day; Doxercalciferol 7.5 mcg/day
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and effectiveness of an investigational drug called doxercalciferol in participants with moderate to severe chronic plaque psoriasis, in comparison with a placebo ("sugar pill"). All study related care was provided including doctor visits, physical exams, laboratory tests and study medication. Total length of participation was 28 weeks.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, placebo-controlled, dose-ranging, parallel group study to evaluate the efficacy and safety of doxercalciferol given orally, once daily for 24 weeks to participants with moderate to severe chronic plaque psoriasis. Participants were randomized and stratified by site and Psoriasis Area Severity Index (PASI) score to one of three active treatment groups or to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Participant had moderate to severe chronic plaque psoriasis defined by a body surface area (BSA) involvement greater than or equal to (>=) 10 percent (%) and plaques with at least a slight elevation above the surrounding normal skin at the Day 1 visit
* Participant had a static Physician's Global Assessment (PGA) of moderate or severe at the Day 1 visit
* Participant had a minimum PASI score of 10 at the Day 1 visit
* Participant was a candidate to receive systemic psoriasis therapy in the opinion of the Investigator
* Participant of childbearing potential, was willing to use an effective contraceptive method throughout the study, which included barrier methods, hormones, or intrauterine devices

Exclusion Criteria:

* Used vitamin D analogues, multivitamin supplements containing greater than (>) 400 international unit (IU) vitamin D, topical retinoids, topical pimecrolimus, and topical tacrolimus within 14 days prior to the Day 1 visit
* Used drugs known to influence serum calcium (such as lithium, digoxin, thiazide diuretics, teriparatide, bisphosphonates, and calcitonin) and multivitamin supplements containing calcium and/or calcium-containing antacids exceeding a total of 1 gram/day within 14 days prior to the Day 1 visit
* Used keratolytics or coal tar (except shampoo containing coal tar or salicylic acid) within 14 days prior to the Day 1 visit
* Used low potency topical corticosteroids (Classes VI and VII), except on the groin, scalp, palms, soles and face, within 14 days prior to the Day 1 visit
* Used medium potency topical corticosteroids (Classes III - V) or high potency topical corticosteroids (Classes I and II) within 14 days prior to the Day 1 visit
* Used systemic retinoids, systemic corticosteroids, methotrexate, cyclosporine, azathioprine, thioguanine or other systemic immunosuppressant agents within 28 days prior to the Day 1 visit
* Used phototherapy, including Ultraviolet B within 14 days or Psoralen plus Ultraviolet A within 28 days prior to the Day 1 visit
* Used a biological agent (including, but not limited to, etanercept, adalimumab, efalizumab, infliximab, or alefacept) within 5 half-lives of the drug prior to the Day 1 visit
* Used systemic antibiotics within 14 days prior to the Day 1 visit. Antibiotic treatment of infections during the Treatment Period was not excluded
* Used investigational drugs within 28 days prior to the Day 1 visit
* Current erythrodermic, guttate, generalized pustular, unstable psoriasis or other chronic active skin conditions that may interfere with the study
* Screening visit laboratory result exceeded the following limits: alanine transaminase (ALT) or aspartate transaminase (AST) >1.5 times the upper limit of normal (ULN); bilirubin >ULN; serum creatinine, calcium, or phosphorus >ULN; spot urine calcium/creatinine ratio >0.4
* History of nephrolithiasis
* Chronic kidney disease as evidenced by a calculated glomerular filtration rate (GFR) less than (<) 60 milliliter/minute/1.73 square meter (mL/min/1.73 m^2) at the screening visit
* Symptomatic coronary or cerebral vascular disease, human immunodeficiency virus, active viral hepatitis, or any other clinically significant, unstable medical condition that would interfere with the completion of the study
* Clinically significant electrocardiogram (EKG) abnormality at screening
* Any evidence of active malignancy except for basal cell carcinoma of the skin. A history of malignancy was not an exclusion
* Active ethanol or drug abuse, excluding tobacco use
* Active severe psychiatric illness that could interfere with the conduct of the study
* Pregnant or breast-feeding women
* Known allergy or hypersensitivity to vitamin D or other ingredients in the study drug formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Hot Springs, Arizona
  - Little Rock, Arkansas
  - Irvine, California
  - Santa Monica, California
  - Alpharetta, Georgia
  - Indianapolis, Indiana
  - Andover, Massachusetts
  - Boston, Massachusetts
  - Troy, Michigan
  - West Bloomfield, Michigan
  - St Louis, Missouri
  - East Windsor, New Jersey
  - Albuquerque, New Mexico
  - Stony Brook, New York
  - Greer, South Carolina
  - Nashville, Tennessee
  - San Antonio, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 centers in the United States of America between April 01, 2008 and June 09, 2009.
Pre-assignment Details: A total of 195 participants were screened of which 84 (43.1%) were screen failures; main reason for screen failure was participant did not qualify for randomization. A total of 111 participants were randomized.
Period: Overall Study
Arm/Group | Placebo | Doxercalciferol 2.5 mcg/Day | Doxercalciferol 5 mcg/Day | Doxercalciferol 7.5 mcg/Day
Started | 27 (Randomized.) | 31 | 28 | 25
Treated | 27 | 31 | 28 | 25
Completed | 14 | 22 | 16 | 13
Not Completed | 13 | 9 | 12 | 12
Not completed — Adverse Event | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 7 | 4
Not completed — Lost to Follow-up | 3 | 3 | 0 | 3
Not completed — Serum Calcium >11.5 milligram/deciliter | 0 | 0 | 0 | 1
Not completed — Worsening of Psoriasis | 4 | 1 | 1 | 4
Not completed — Undefined | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Doxercalciferol 2.5 mcg/Day | Doxercalciferol 5 mcg/Day | Doxercalciferol 7.5 mcg/Day | Total
Number analyzed (Participants) | 27 | 31 | 28 | 25 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (11.9) | 40.5 (12.4) | 49.9 (12.6) | 44.2 (16.3) | 44.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 10 | 10 | 40
  Male | 18 | 20 | 18 | 15 | 71
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 2 | 3 | 0 | 2 | 7
  White | 22 | 27 | 26 | 22 | 97
  Multiple | 0 | 0 | 1 | 1 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Body mass index was calculated by dividing body weight (kilogram) by the height (meters) squared.
  kilogram per square meter (kg/m^2) | 32.4 (7.5) | 33.9 (8.3) | 30.1 (6.5) | 32.7 (9.8) | 32.3 (8.1)
Week 0/Day 1 Psoriasis Area Severity Index (PASI) Score [Number; unit: participants] — PASI score: range: 0 (no disease) to 72 (maximal disease). Body was divided into head (h), trunk (t), upper (u) and lower (l) extremities. For each section, percent area of skin involved (A) was estimated: 1 (less than [<] 10%) to 6 (90% - 100%), and severity was estimated by clinical signs: (erythema [E], induration [I], and desquamation [D]) on a scale: 0=no symptoms, 4=very marked. PASI score= 0.1 (E[h] + I[h] + D[h]) A[h] + 0.2 (E[u] + I[u] + D[u]) A[u] + 0.3 (E[t] + I[t] + D[t]) A[t] + 0.4 (E[l] + l[I] + D[l]) A[l]. Number of participants with PASI score <=16 and >16 are reported.
  participants
    Less Than or Equal to (<=) 16 | 15 | 16 | 16 | 14 | 61
    Greater Than (>) 16 | 12 | 15 | 12 | 11 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 50 Percent (%) Reduction in Psoriasis Area Severity Index (PASI) Score at Week 12 or Early Termination
Description: PASI score: range: 0 (no disease) to 72 (maximal disease). Body was divided into head (h), trunk (t), upper (u) and lower (l) extremities. For each section, percent area of skin involved (A) was estimated: 1 (<10%) to 6 (90% - 100%), and severity was estimated by clinical signs: (erythema [E], induration [I], and desquamation [D]) on a scale: 0=no symptoms, 4=very marked. PASI score= 0.1 (E[h] + I[h] + D[h]) A[h] + 0.2 (E[u] + I[u] + D[u]) A[u] + 0.3 (E[t] + I[t] + D[t]) A[t] + 0.4 (E[l] + l[I] + D[l]) A[l].
Time Frame: Week 12 or Early Termination
Population: The Full Analysis Set (FAS) included all safety set-evaluable participants with at least one post-baseline PASI assessment after the date of first dose in the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Doxercalciferol 2.5 mcg/Day | Doxercalciferol 5 mcg/Day | Doxercalciferol 7.5 mcg/Day
Number analyzed (Participants) | 25 | 30 | 28 | 25
percentage of participants | 20.0 | 20.0 | 17.9 | 20.0
Statistical Analysis 1: Comparison: Placebo vs Doxercalciferol 2.5 mcg/Day; Estimate of the log odds, relative to the Placebo, in participants with at least 50 % reduction in PASI score at Week 12 or early termination was analyzed using exact logistic regression model adjusted for site and baseline PASI strata (<=16, >16); Test type: Superiority or Other; p = 1.000, Regression, Exact Logistic — The p-value was not adjusted for multiple comparisons or a prior significance threshold; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.17 to 4.22]
Statistical Analysis 2: Comparison: Placebo vs Doxercalciferol 5 mcg/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.992, Regression, Exact Logistic — The p-value was not adjusted for multiple comparisons or a prior significance threshold; Odds Ratio (OR) = 0.76, 95% CI [0.13 to 4.14]
Statistical Analysis 3: Comparison: Placebo vs Doxercalciferol 7.5 mcg/Day; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.000, Regression, Exact Logistic — The p-value was not adjusted for multiple comparisons or a prior significance threshold; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.15 to 4.59]

2. Secondary Outcome: Percentage of Participants With at Least 50 Percent (%) Reduction in Psoriasis Area Severity Index (PASI) Score at Week 24 or Early Termination
Description: as for outcome 1
Time Frame: Week 24 or Early Termination
Population: FAS included all safety set-evaluable participants with at least one post-baseline PASI assessment after the date of first dose in the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Doxercalciferol 2.5 mcg/Day | Doxercalciferol 5 mcg/Day | Doxercalciferol 7.5 mcg/Day
Number analyzed (Participants) | 25 | 30 | 28 | 25
percentage of participants | 36.0 | 20.0 | 21.4 | 32.0

3. Secondary Outcome: Percentage of Participants With Static Physician's Global Assessment (PGA) Score of Clear or Almost Clear at Week 12, 24 or Early Termination
Description: Static PGA of psoriasis is scored on a 5-point scale (0 = clear to 4 = severe), reflecting a global consideration of the erythema, induration and scaling across all psoriatic lesions. Clear (erythema: no, scale: no, induration: no thickness); Almost Clear (erythema: light pink, scale: fine scale, induration: barely palpable); Mild (erythema: light red, scale: coarse scale on most lesions, induration: slight but visible elevation, indistinct edges); Moderate (erythema: red, scale: coarse adherent scale predominates, induration: moderate elevation with edges); and Severe (erythema: dark red to purple, scale: thickened adherent scale, induration: marked thickness distinct and pronounced edges). Percentage of participants with static PGA score of clear or almost clear are reported.
Time Frame: Week 12 or Early Termination, Week 24 or Early Termination
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Doxercalciferol 2.5 mcg/Day | Doxercalciferol 5 mcg/Day | Doxercalciferol 7.5 mcg/Day
Number analyzed (Participants) | 25 | 30 | 28 | 25
percentage of participants
  Week 12 or Early Termination | 0 | 6.7 | 3.6 | 0
  Week 24 or Early Termination | 8.0 | 3.3 | 10.7 | 16.0

ADVERSE EVENTS:
Time Frame: Reported adverse events include the treatment-emergent events starting on or after the day of study drug administration up to Week 28 or Early Termination
Description: Analysis was performed on Safety Set, defined as all randomized participants who received at least 1 dose of study medication. In the event a single participant experienced both serious and non-serious forms of the same adverse events, the individual was included in the numerator (number of participants affected) of each adverse event table.
Arm/Group | Placebo | Doxercalciferol 2.5 mcg/Day | Doxercalciferol 5 mcg/Day | Doxercalciferol 7.5 mcg/Day
Serious Adverse Events (participants affected / at risk) | 0/27 | 2/31 | 1/28 | 1/25
Other Adverse Events (participants affected / at risk) | 8/27 | 16/31 | 14/28 | 5/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Doxercalciferol 2.5 mcg/Day (N=31) | Doxercalciferol 5 mcg/Day (N=28) | Doxercalciferol 7.5 mcg/Day (N=25)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Doxercalciferol 2.5 mcg/Day (N=31) | Doxercalciferol 5 mcg/Day (N=28) | Doxercalciferol 7.5 mcg/Day (N=25)
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 5 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Citric acid urine decreased (Investigations) | 0 | 0 | 2 | 0
Urine electrolytes increased (Investigations) | 0 | 0 | 2 | 0
Urine uric acid increased (Investigations) | 0 | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.